CLINICAL TRIAL: NCT02135523
Title: The Efficacy of Involved-field Radiation Therapy for Residual or Locoregionally Recurrent Epithelial Ovarian Cancer After Definitive Treatment; Multi-institutional Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2013-0896
Record Dates: First submitted 2014-04-23; First posted 2014-05-12 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Ovarian Cancer (Epithelial)
Keywords: ovarian cancer; involved-field radiation therapy; progression free survival
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm: involved-field radiation therapy group (Experimental)
  Interventions: Radiation: involved-field radiation therapy

INTERVENTIONS:
Radiation: involved-field radiation therapy — Participants will receive involved-field radiotherapy (external beam radiotherapy or brachytherapy) over 45Gy for residual or locoregionally recurrent epithelial ovarian cancer after definitive treatment. Patients will be treated with 1.8-2.0Gy fraction, five times per week. It starts 2 weeks later of chemotherapy.

SUMMARY:
1. Title: The efficacy of involved-field radiation therapy for residual or locoregionally recurrent epithelial ovarian cancer after definitive treatment; Multi-institutional phase 2 clinical trial
2. Study period: 2014.04~2018.04
3. Objective: To determine whether involved-field radiation therapy will prove to be improve 2-year progression free survival for residual or locoregionally recurrent epithelial ovarian cancer patients after definitive treatment.
4. Patient Selection: primary epithelial ovarian cancer (Required sample size: 70)
5. Planned number of patients

   * YUHS database have 149 FIGO stage III patients treated with debulking surgery and adjuvant platinum-based chemotherapy 2.
   * Of these patients, 90 patients experienced locoregional failures, and then the investigators selected 44 patients who could be treated effectively with IFRT based on MDACC suggestion.
   * Median interval to failure was 9 months in these patients

     * Hypothesis; IFRT reduces 44% hazard of progression compared with patients without IFRT
     * Sample size; two-sided, accrual time = 24 mo, f/u time= 36 mo. α= 0.05, power = 0.80 Null progression-free median survival = 9 mo Alt progression-free median survival = 16 mo Calculated sample number = total 27 patients Drop rate = 10% • Total sample number = 30 patients Estimated Enrollment : 30 participants

Drop rate = 10%

* Total sample number = 70 patients 6. Radiation therapy: Participants will receive involved-field radiotherapy (external beam radiotherapy or brachytherapy) over 45Gy with 1.8-2.0 Gy fraction, five times per week for residual or locoregionally recurrent epithelial ovarian cancer after definitive treatment
* Target volume

  * directed to gross disease plus a high-risk clinical target volume (CTV) that included the postoperative bed or the prechemotherapy extent of disease with a 1- to 1.5-cm margin, excluding uninvolved clinical structures
  * Additional CTVs were designated according to the risks of microscopic disease spread, proximity to critical structures, and other risk factors for complications.
  * Nodal CTVs included grossly involved lymph node sites, extending to cover adjacent uninvolved regions.
* Modality; 3-dimensional conformal RT including electron, intensity-modulated RT, proton beam RT 7. Patient assessment: Participants will be followed at 1, 3, 6, 12, 18 and 24 month after radiation therapy 8. Key words: ovarian cancer, involved-field radiation therapy, progression free survival

ELIGIBILITY:
Inclusion Criteria:

1. age> 19 years
2. ECOG performance status 0-1
3. pathologically confirmed malignant epithelial ovarian cancer
4. surgically removal of tumor including both ovary resection, total hysterectomy, lymph node and mesentery
5. at least on of the following: consolidation therapy for grossly negative condition prior large tumor after surgery and adjuvant chemotherapy, residual tumor after adjuvant or salvage chemotherapy, local recurrent tumor after adjuvant or salvage chemotherapy, consolidation therapy after surgical removal of recurrent tumor

Exclusion Criteria:

1. diffuse peritoneal seeding
2. brain or bone metastasis
3. prior invasive malignancy (except controlled skin cancer, carcinoma in situ of the cervix and early thyroid and gastric cancer) unless disease free for a minimum of 5 years prior to study entry
4. serious underlying medical disease
5. not providing informed consent

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-02-06 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Two-year progression free survival(PFS) after involved-field radiation therapy | Participants will be followed for 2 year after radiation therapy
  To determine whether involved-field radiation therapy will prove to be improved 2-year progression free survival for residual or locoregionally recurrent epithelial ovarian cancer patients after definitive treatment.

SECONDARY OUTCOMES:
overall survival | Participants will be followed at 1, 3, 6, 12, 18 and 24 month after radiation therapy
chemotherapy-free survival | Participants will be followed at 1, 3, 6, 12, 18 and 24 month after radiation therapy
in-field disease control | Participants will be followed at 1, 3, 6, 12, 18 and 24 month after radiation therapy
serious adverse event | Participants will be followed at 1, 3, 6, 12, 18 and 24 month after radiation therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Korea, South Korea